CLINICAL TRIAL: NCT01019824
Title: A Phase III Study to Assess the Efficacy and Safety of Ralfinamide.
Brief Title: Efficacy and Safety of Ralfinamide in Patients With Chronic Neuropathic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Collaborators: Parexel (Industry); CliniRx (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NW-1029/01-08; EudraCT Nr.: 2008-006176-30 (Other: EMEA)
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Pain
Keywords: nerve compression; compression radiculopathy; post-traumatic/post-surgical lumbar radiculopathy
MeSH Terms: conditions — Pain; Neuroma | interventions — Ralfinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose (Experimental): 160 mg dose
  Interventions: Drug: Ralfinamide
- High Dose (Experimental): 320 mg dose
  Interventions: Drug: Ralfinamide
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Ralfinamide

INTERVENTIONS:
Drug: Ralfinamide — Ralfinamide Oral Tablets, 160 or 320 mg per day

SUMMARY:
The aim of the study is to determine if an experimental drug, ralfinamide, relieves your neuropathic low back pain, and if it demonstrates superiority to placebo, a "dummy" or sugar pill that contains no active medication. Ralfinamide, given as either 160 mg/day or 320 mg/day, taken in a divided dose twice-a-day, will be compared with placebo. If you are randomly (by chance) selected to receive placebo, you will receive this medication throughout the treatment period of the study. Data from this study will provide essential information for choosing the doses of ralfinamide to be used in the treatment of this type of pain and potentially other types of pain.

DETAILED DESCRIPTION:
Ralfinamide has been shown to be an effective analgesic in a number of animal models of neuropathic pain. These observed effects of ralfinamide may have been achieved by targeting both hyperactivity of peripheral sensory neurons, through voltage-dependent, Na+-channel blockade [Stummann et al., 2005] and Ca++-channel blockade, and sensitization of central neurons, through NMDA-receptor modulation.

Evidence of efficacy in mixed peripheral neuropathic pain syndromes has been demonstrated in Study 001 [Anand et al., 2008]. In particular patients with neuropathic pain due to nerve compression (e.g., compression radiculopathy, lumbar spinal stenosis, sciatic nerve compression, spinal root compression, intercostal neuralgia) showed response to ralfinamide treatment. In this sub-population, statistically significant improvements in severity of pain, as measured on the VAS and 11-point Likert scales, as well as a greater proportion of patients meeting "responder" criteria, compared to the placebo group, were noted with ralfinamide treatment. Similarly, patients in the study classified as having neuropathic low back pain also showed significant benefit from treatment with ralfinamide; therefore, the focus of the current study is on this indication.

The current study will evaluate the safety, tolerability and analgesic efficacy of ralfinamide in patients with chronic neuropathic low back pain due to nerve compression, i.e., compression radiculopathy or post-traumatic/post-surgical lumbar radiculopathy. It should also be noted that no current drug therapy has global regulatory approval for treating this type of chronic neuropathic low back pain; therefore, should ralfinamide prove effective in this patient population, it would be satisfying an unmet medical need.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for enrolment into the study:

  1. Patient presents in the physical/neurological examination with low back pain with or without radiation into the lower limb that must display a topography compatible with the L1 to S1 territory and/or respective sensory or motoric impairments.
  2. Patient must have chronic neuropathic low back pain with a minimum intensity of "40 mm" (moderate) or greater on the Visual Analogue Scale (VAS; 100-mm) at screening, and an average of "40 mm" or more at baseline (based on prior 7 days).
  3. The onset of pain has occurred at least three months, but not longer than 3 years, prior to the screening visit, as assessed by the investigator in the patient's medical history.
  4. Patient is affected by current neuropathic pain (pain provoked by a lesion of the peripheral nervous system). The diagnosis should be made by a neurologist/anaesthesiologist/pain specialist and based on history, clinical evaluation and/or laboratory findings (rule out systemic cause, e.g., hypothyroidism, rheumatoid arthritis, nephropathy, diabetes [MNSI score >2]) in accordance with the taxonomy of the diagnostic criteria documented in the International Association for the Study of Pain (IASP) Classification of Chronic Pain. A neurological disease must be directly correlated with pain, including pain due to spinal root compression.

     If radiologic data supporting the diagnosis had been obtained previously it should be documented in the patient's records. In case radiologic examinations are not available, the Investigator should consider performing these examinations, if necessary to support the diagnosis, during the screening phase.
  5. Patient has one of the following causes of neuropathic low back pain: Non-cancer lumbar pain due to compression radiculopathy or post-traumatic/post-surgical lumbar radiculopathy.
  6. Patient's low back pain has a clear neuropathic component, as indicated by a rating on the Pain Detect Questionnaire (PD-Q) of greater than 18.
  7. Patient is 18-85 years of age, inclusive.
  8. Patient is willing and able to understand and sign an approved Informed Consent Form.

Exclusion Criteria:

* 1. Females who are pregnant or lactating, or of childbearing potential, defined as follows: surgically sterilized for less than one year; aged ≥ 50 years and post-menopausal condition started less than 24 months prior to the screening visit; or aged < 50 years and post-menopausal condition started less than 24 months prior, and/or post-menopausal status has not been confirmed by determination of the serum levels of FSH and 17-β estradiol; or fecund and not practicing double contraception method (e.g., hormonal contraceptive plus barrier method).

  2. Patients with any other cause of peripheral or central neuropathic pain (including psychogenic and nociceptive pain), pain due to metabolic (including diabetes; MNSI score > 2) infectious or proliferative diseases, or pain due to any condition that is as severe as the neuropathic pain.

  3. Patients with a history of migrating pain and former mononeuropathy or neuralgias in other anatomical territories.

  4. Patients with severe trophic changes, severe swelling, joint deformities or stiff joint with limited passive movement, or patients who may be candidates for back surgery within 52 weeks after baseline.

  5. History or current diagnosis of positive test for Hepatitis B or C (unless vaccinated).

  6. Clinically significant, uncontrolled gastrointestinal, renal, hepatic, endocrine, pulmonary or cardiovascular disease (including non well-controlled hypertension), asthma, uncompensated chronic obstructive pulmonary disease (COPD), severe uncontrolled diabetes (HbA1c > 10.0).

  7. Second- or third-degree atrioventricular block or sick sinus syndrome, uncontrolled atrial fibrillation, severe or unstable angina, congestive heart failure, myocardial infarction within 3 months of the screening visit, significant ECG abnormalities or QTc ≥ 450 msec (males) or ≥ 470 msec (females), where QTc is based on Bazett's correction method.

  8. Concomitant disease likely to interfere with the study drug (e.g. capable of altering absorption, metabolism or elimination of drugs).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2009-03-20 (Actual); Primary Completion 2010-05-11 (Actual); Study Completion 2011-08-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be the change from baseline in the mean weekly pain score (11-point Likert scale). | The primary efficacy endpoint will analyze the change from baseline to Week 12 of the mean weekly pain score

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Rossetti, MD, Study Director — Newron Pharmaceuticals SPA
Locations (1):
- Parexel, London, England, United Kingdom